CLINICAL TRIAL: NCT05041348
Title: Affiliated Hospital of Qingdao University
Brief Title: Metabonomic of Patients With Hepatitis B Cirrhosis Complicated With Sarcopenia.
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: QYFYWZLL26461
Record Dates: First submitted 2021-07-15; First posted 2021-09-13 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Sarcopenia
Keywords: Hepatitis B virus-related liver cirrhosis; muscle mass loss; metabolites
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- liver cirrhosis patients with muscle mass loss: The diagnosis of cirrhosis was made based on the combination of clinical and laboratory features or by liver histopathology. Skeletal muscle mass index (SMI), which was the ratio of lean tissue area to body height. Muscle mass loss was defined as an SMI less than 46.96 cm²/m² for males and less than 32.46 cm²/m² for females
  Interventions: Diagnostic Test: CT at the level of the third lumbar vertebra (L3)
- liver cirrhosis patients with normal muscle mass: Skeletal muscle mass index (SMI) was not decreased in this group.
  Interventions: Diagnostic Test: CT at the level of the third lumbar vertebra (L3)
- healthy group: People in healthy control group were excluded metabolic diseases (including diabetes, thyroid disorder, and so on) and other chronic diseases, according to their ultrasound and laboratory assessment.

INTERVENTIONS:
Diagnostic Test: CT at the level of the third lumbar vertebra (L3) — Muscle mass loss was defined as an skeletal muscle mass index (SMI) less than 46.96 cm²/m² for males and less than 32.46 cm²/m² for females
  Groups: liver cirrhosis patients with muscle mass loss; liver cirrhosis patients with normal muscle mass

SUMMARY:
Sarcopenia is a common complication in liver cirrhosis patients and has been confirmed that associated with poor prognosis. China has the world's largest burden of hepatitis B virus-related liver cirrhosis (HBV-related liver cirrhosis). However, the relationship between HBV-related liver cirrhosis patients with muscle mass loss and normal muscle mass is remain largely unknown. Our study aimed to reveal the metabolic profile and identify potential biomarkers of muscle mass loss in HBV-related liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. the diagnostic criteria for decompensation of liver cirrhosis of chronic viral hepatitis B formulated according to the Guidelines for Diagnosis and Treatment of Liver Cirrhosis issued by the Chinese Society of Hepatology in 2019
2. The diagnosis of muscle mass loss conforms to SMI less than 46.96 cm²/m² for males and less than 32.46 cm²/m² for females
3. Patients aged between 18 and 60 years old
4. Patients with no history of drinking or abstinence for more than 1 year
5. Voluntary participants with informed consent

Exclusion Criteria:

1) the etiology of cirrhosis without hepatitis B virus (HBV), such as cirrhosis, alcoholic cirrhosis, autoimmune cirrhosis, and so on; 2) the age of patients over 60 years old; 3) patients with acute, chronic and acute liver failure; 4) other diseases which can lead to the secondary muscle depletion, such as chronic disease in heart, lung, kidney, brain, and malignant tumor; 5) neurodegenerative diseases or muscle degenerative diseases; 6) perioperative patients; 7) patients without CT scan within 3 months; 8) patients who have exercise habits with the Physical Activity Rating Scale-3 (PARS-3) > 19 points

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with HBV-related liver cirrhosis were recruited between August 2021 and June 2022 at the Affiliated hospital of Qingdao University. All of the patients are in the decompensation stage of hepatitis B cirrhosis and divided them into two groups. One group is named cirrhosis with muscle mass loss, the other group is named liver cirrhosis with normal muscle mass. People in healthy control group were excluded metabolic diseases. Each group of patients is about 20.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
amino acids metabolism | 2021.09.01-2022.08.01
  Arginine biosynthesis, Phenylalanine, tyrosine and tryptophan biosynthesis were the enrichment pathway in two groups.
central carbon metabolism | 2021.09.01-2022.08.01
  D-fructose-6-phosphate,L-glutamic acid, and Fumaric acid were selected as differential metabolites in pathway of central carbon metabolism.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, China

IPD SHARING:
Plan to Share IPD: No